CLINICAL TRIAL: NCT00711724
Title: Comparison of Self and Clinician Administered Rating Scales in Patients With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Comparison of Self and Clinician Administered Rating Scales in Patients With ADHD
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Paul Hammerness, MD, Massachusetts General Hospital
Other Study IDs: 2007-P-000911
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2010-06

CONDITIONS: Attention-Deficit/Hyperactivity Disorder (ADHD)
Keywords: Attention Deficit Hyperactivity Disorder (ADHD); Adolescent
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MGH 1: Adolescents with Attention Deficit Hyperactivity Disorder (ADHD)

SUMMARY:
The primary objective is to establish the concurrent validity of the clinician administered Attention Deficit Hyperactivity Disorder-Rating Scale (ADHD-RS) and the patient administered Attention Deficit Hyperactivity Disorder Self Report Scale (ASRS) v1.1 Symptom Checklist.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHD
* Age 13-65* *Parental consent and patient's assent will be obtained for minors participating in this protocol (only adolescents aged 13-18 yrs old will be included in the MGH site)

Exclusion Criteria:

* Inability to reliably report ADHD symptoms at the discretion of the investigator

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents diagnosed with Attention Deficit Hyperactivity Disorder (ADHD) who are enrolled in the study Protocol 2003-P-001313: "Prevention of Cigarette Smoking in ADHD Youth with CONCERTA."
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The ADHD-RS and ASRS v1.1 Symptom Checklist scales | Weeks 1, 2, 3, 4, 5, 6, 7, or 8

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hammerness, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States

REFERENCES:
- See also: Related Info — http://massgeneral.org/pediatricpsych/home.html